CLINICAL TRIAL: NCT00709319
Title: Evaluation of Vitrectomy for Diabetic Macular Edema Study
Brief Title: Evaluation of Vitrectomy for Diabetic Macular Edema
Acronym: Vitrectomy-D
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NEI-125; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetic retinopathy; Diabetic macular edema; dme; vitrectomy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: Subjects vitreomacular traction, visual acuity 20/63 to 20/400, retinal thickness >300 microns in the central subfield on OCT, and cataract extraction not being performed in conjunction with vitrectomy.

SUMMARY:
The study is designed as a prospective cohort study to assess changes in visual acuity and retinal thickening and surgical complications in subjects undergoing vitrectomy for diabetic macular edema.

The study also aims to identify subgroups in which there appears to be a benefit of vitrectomy and subgroups in which vitrectomy does not appear to be beneficial and to obtain data that can be used to plan a randomized trial.

Subject will be followed through 2 years, with a primary outcome at 6 months post vitrectomy surgery. The vitrectomy procedure will be performed based on the investigators usual care and is not considered part of the research although the procedure performed will be collected.

DETAILED DESCRIPTION:
Study Design The study is designed as a prospective cohort study. A randomized trial design was considered but rejected after deciding that there was insufficient equipoise on the part of the investigator group to randomize eyes with DME and vitreal traction to surgery or no surgery (thus eyes which potentially may benefit most from vitrectomy would not be included), and there was insufficient information available on the natural course or surgical outcomes of eyes with DME but without significant traction.

A cohort study provides the opportunity to collect data prospectively using a standardized protocol to assess the potential benefits and risks of vitrectomy. The results can be used to determine whether proceeding with a randomized trial has merit and what the design of the trial should be. If a randomized trial is to be conducted, the results plus the cohort study experience can be used to help design the protocol.

Study Objectives

1. To provide information on the following outcomes in eyes with Diabetic Macular Edema (DME) that undergo vitrectomy: visual acuity, retinal thickening, resolution of traction (if present), surgical complications.
2. To identify subgroups in which there appears to be a benefit of vitrectomy and subgroups in which vitrectomy does not appear to be beneficial.
3. To obtain data that can be used to plan a randomized trial.

B. Intervention Vitrectomy performed by the investigator's usual routine.

C. Duration of Follow-Up: Two years

D. Follow-up Visit Schedule Study visits for data collection at 3 and 6 months then 1, and 2 years. Additional visits follow investigator's usual routine.

E. Rationale:

There are at least two avenues of investigation that support the theoretical value of vitrectomy for the treatment of DME, based on (1) vitrectomy for the relief of traction on the macula and (2) vitrectomy to improve oxygenation of the macula leading to decreased permeability with subsequent resolution or decrease in DME.

Vitrectomy to relieve biomechanical traction on the macula has been reported widely. Schepens and coworkers discussed the role of the vitreous and vitreomacular traction in cystoid macular edema in 1984. Nasrallah et al observed in 1988 the resolution of diabetic macular edema in individuals with spontaneous separation of the vitreous gel from the retina. In 1992, Lewis and coworkers reported success with vitrectomy and peeling of a "thickened hyaloid membrane" in eyes with DME that had this anatomical feature. Since this report of a nonrandomized retrospective case series, other authors have prospectively analyzed their series and supported the concept that relief of clear-cut anteroposterior traction, usually in the setting of an epiretinal membrane complex and associated vitreous adherence, may ameliorate macular thickening and edema in DME. Evaluation of these individuals and documentation of pre and postoperative characteristics have been rendered vastly more objective by ocular coherence tomography and the Retina Thickness Analyzer. Series using optical coherence tomography (OCT) to image cases where vitreomacular traction is observed and in some cases treated, has confirmed the clinical impression of mechanical forces at work on the posterior retina and has documented the anatomic improvement with surgery. How and in which cases OCT could refine our ability to diagnose and define clinically important anatomical features or relationships has not been investigated. As Kaiser and coworkers have documented, the OCT findings in the cases that have thus far come to vitrectomy in these situations support a conclusion that the disease process has progressed very far and in many cases the individuals have actual traction retinal detachments in their maculae. These severe cases are the exception in the spectrum of DME: most cases of macular edema have no obvious vitreomacular traction, but this factor has not been investigated adequately with our newer and more sophisticated imaging techniques. It is possible that subclinical traction on the macula exists in a large number of individuals with diabetes, whose internal limiting membranes at the vitreomacular interface often have a thickened, hypercellular appearance and whose vitreous gels, gradually contracting over many years, may exert subclinical but significant traction on the compromised diabetic macular vascular bed.

The other line of reasoning and prior research that supports the possibility that vitrectomy would help DME is that articulated by Steffanson and others indicating that posterior segment oxygenation improves after vitrectomy. Using oxygen sensors on the retinal surface, these investigators have shown that retinal oxygen tensions increase after the vitreous gel is removed and the posterior segment becomes perfused by relatively oxygen-rich aqueous humor. Supporting this conclusion is the additional observation that retinal vessels decrease in caliber after vitrectomy, presumably in response to the improvement in hypoxia, although confounding factors that could contribute to this decrease, such as the addition of endolaser retinal photocoagulation, have not been ruled out. Numerous lines of investigation have elucidated factors producing permeability in retinal blood vessels. One of the most central of these factors is Vascular Endothelial Growth factor (VEGF), formerly known as Vascular Permeability Factor (VPF). VEGF is known to be upregulated by hypoxia, and downregulated by increased oxygenation. The speculated sequence of events in which vitrectomy produces improved oxygenation of the posterior segment, leading to downregulation of VEGF, leading to decreased vasopermeability, resulting in reduced macular thickening, is a plausible one. More rapid clearing of growth factors in the vitrectomized eye has also been postulated as a potential mechanism for this response.

See full protocol at drcr.net for list of references

ELIGIBILITY:
Subject-level Inclusion Criteria

To be eligible, the following inclusion criteria (1-3) must be met:

1. Age >= 18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. Able and willing to provide informed consent.

   Subject-level Exclusion Criteria

   A patient is not eligible if any of the following exclusion criteria (4-6) are present:
4. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
5. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first year of the study.
6. Blood pressure >180/110 (systolic above 180 OR diastolic above 110).

Study Eye Criteria

To be a study eye, all of the inclusion criteria (a-e) and none of the exclusion criteria (f-m) listed below must be met. A patient can have only one study eye. If both eyes are eligible and undergoing vitrectomy, the first eye having surgery will be the study eye.

The eligibility criteria for a study eye are as follows:

Inclusion

1. Vitrectomy being performed as treatment for DME.
2. E-ETDRS visual acuity 20/800 or better (E-ETDRS visual acuity score >= 3 letters).
3. Definite retinal thickening due to diabetic macular edema based on clinical exam involving the center of the macula.
4. Presence of vitreomacular traction associated with macular edema OR edema is felt to be too diffuse to respond to focal or grid laser OR edema judged to be inadequately responsive to previous treatment(s) and unlikely to benefit from further focal photocoagulation.
5. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs.

   Exclusion
6. Macular edema is considered to be due to a cause other than diabetic macular edema.
7. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary abnormalities, subfoveal hard exudates, fibrous metaplasia, nonretinal condition).
8. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, post-surgical cystoid macular edema, etc.).
9. History of retinal macular photocoagulation, intravitreal corticosteroids, or other treatment for DME within 3.5 months prior to enrollment.
10. History of peripheral scatter photocoagulation within 4 months prior to enrollment or anticipated need within the 4 months following enrollment.
11. History of prior pars plana vitrectomy.
12. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following enrollment.
13. History of YAG capsulotomy performed within 2 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with diabetic macular edema
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia A. Haller, M.D., Study Chair — Wills Eye Institute
Locations (48):
- United States (48):
  - University of California, Irvine, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - West Coast Retina Medical Group, Inc., San Francisco, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Retina Associates of Hawaii, Inc., Honolulu, Hawaii
  - Retina Consultants of Hawaii, Inc., ‘Aiea, Hawaii
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Associated Retina Consultants, Williamsburg, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - Retina Consultants, PLLC, Slingerlands, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Charlotte Eye Ear Nose and Throat Assoc, PA, Charlotte, North Carolina
  - Horizon Eye Care, PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Charles A. Garcia, PA & Associates, Houston, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin

REFERENCES:
- [Background] Diabetic Retinopathy Clinical Research Network Writing Committee; Haller JA, Qin H, Apte RS, Beck RR, Bressler NM, Browning DJ, Danis RP, Glassman AR, Googe JM, Kollman C, Lauer AK, Peters MA, Stockman ME. Vitrectomy outcomes in eyes with diabetic macular edema and vitreomacular traction. Ophthalmology. 2010 Jun;117(6):1087-1093.e3. doi: 10.1016/j.ophtha.2009.10.040. Epub 2010 Mar 17. PMID 20299105
- [Background] Flaxel CJ, Edwards AR, Aiello LP, Arrigg PG, Beck RW, Bressler NM, Bressler SB, Ferris FL 3rd, Gupta SK, Haller JA, Lazarus HS, Qin H. Factors associated with visual acuity outcomes after vitrectomy for diabetic macular edema: diabetic retinopathy clinical research network. Retina. 2010 Oct;30(9):1488-95. doi: 10.1097/IAE.0b013e3181e7974f. PMID 20924264
- [Derived] Gangaputra S, Almukhtar T, Glassman AR, Aiello LP, Bressler N, Bressler SB, Danis RP, Davis MD; Diabetic Retinopathy Clinical Research Network. Comparison of film and digital fundus photographs in eyes of individuals with diabetes mellitus. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6168-73. doi: 10.1167/iovs.11-7321. PMID 21571677

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Macular Edema and Vitreomacular Traction: The primary cohort included 87 eyes (one eye per participant) with DME and vitreomacular traction based on investigator's evaluation, visual acuity 20/63-20/400, optical coherence tomography (OCT) central subfield greater than 300 microns and no concomitant cataract extraction at the time of vitrectomy.Surgery was performed according to the investigator's usual routine. Follow-up visits were performed after 3 months, 6 months (primary end point), and 1 year.
Period: Overall Study
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Started | 87
Completed | 81
Not Completed | 6
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Diabetic Macular Edema and Vitreomacular Traction: The primary cohort included 87 eyes with DME and vitreomacular traction based on investigator's evaluation, visual acuity 20/63-20/400, optical coherence tomography (OCT) central subfield greater than 300 microns and no concomitant cataract extraction at the time of vitrectomy.Surgery was performed according to the investigator's usual routine. Follow-up visits were performed after 3 months, 6 months (primary end point), and 1 year. Only one eye per participant could be enrolled.
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 66 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 48
Race/Ethnicity, Customized [Number; unit: participants]
  White | 69
  African American | 7
  Hispanic | 5
  Other | 6
Surgery characteristic: Focal/grid laser to diabetic macular edema used [Number; unit: Participants]
  Yes | 4
  No | 83
Surgery characteristic: Panretinal photocoagulation, history of prior use [Number; unit: Participants]
  Yes | 16
  No | 71
Indocyanine green used to improve visualization [Number; unit: Participants]
  Yes | 24
  No | 63
Diabetes Type [Number; unit: Participants]
  Type 1 | 14
  Type 2 | 73
Epiretinal Membranes Present [Number; unit: Participants] — Assessment based on investigators assessment at enrollment.
  Participants
    No | 21
    Probable | 19
    Definite | 43
    Can not deterimine | 4
Lens Status [Number; unit: Participants]
  Phakic | 37
  Pseudophakic/aphakic | 50
Prior Scatter Photocoagulation [Number; unit: Participants]
  Yes | 39
  No | 48
Prior Treatment for Diabetic Macular Edema [Number; unit: Participants]
  Yes | 51
  No | 36
Reasons for Vitrectomy: Vitreomacular interface abnormality [Number; unit: Participants] | 87
Retinopathy Severity [Number; unit: Participants]
  Microaneurysms only | 1
  Mild/moderate nonproliferative diabetic retinopath | 6
  Moderate/severe nonproliferative diabetic retinopa | 14
  Severe nonproliferative diabetic retinopathy | 4
  Proliferative diabetic retinopathy | 51
  Retinal volume not obtained | 11
Status of the Vitreous [Number; unit: Participants] — Status determined from investigators observations at enrollment.
  Participants
    Attached | 49
    Partially Attached | 28
    Detached | 5
    Uncertain | 5
Triamcinolone acetonide used to improve visualization [Number; unit: Participants] — Same subjects could be listed for multiple categories
  Participants
    Yes | 30
    No | 57
Surgical Characteristic: Internal Limiting Membrane Removed [Number; unit: Participants]
  Yes | 47
  No | 40
Surgical Characteristic: Focal to grid breaks Laser Used [Number; unit: Participants]
  Yes | 14
  No | 73
Surgical Characteristic: Vitrectomy System [Number; unit: Participants]
  19/20 gauge | 35
  25 gauge | 43
  23 gauge | 9
Surgical Charachteristic:Epiretinal membrane peeled [Number; unit: Participants]
  Yes | 53
  No | 34
Central Subfield Thickness [Median (Inter-Quartile Range); unit: Microns] | 491 [356 to 586]
Duration of Diabetes [Median (Inter-Quartile Range); unit: Years] | 20 [12 to 25]
Electronic-Early Treatment Diabetic Retinopathy Study Visual Acuity Letter Score [Median (Inter-Quartile Range); unit: Number on a Scale] — Visual Acuity Letter Score Scale: 100 being the best and 0 the worst
  Number on a Scale | 52 [41 to 58]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percent] | 7.1 [6.7 to 7.9]
Retinal Volume [Median (Inter-Quartile Range); unit: mm3] | 9.2 [8.5 to 11.8]
Reasons for Vitrectomy: Unresponsive to other therapies [Number; unit: Participants]
  Yes | 27
  No | 60
Trypan blue used to improve visualization [Number; unit: Participants]
  Yes | 2
  No | 85
Surgery characteristic: Panretinal photocoagulation, with none used prior [Number; unit: Participants]
  Yes | 19
  No | 68
Surgery characteristic: Laser used with endoprobe [Number; unit: Participants]
  Yes | 21
  No | 66
Surgery characteristic: Laser used with indirect ophthalmoscope [Number; unit: Participants]
  Yes | 7
  No | 80
Surgery characteristic: Scatter laser over peripheral schisis or barrier laser used [Number; unit: Participants]
  Yes | 4
  No | 83

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Change in best correct visual acuity letter score from baseline to six months as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best value on the scale 97, worst 0.
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
Units on a scale | 52 [42 to 64]

2. Primary Outcome: Change in Optical Coherence Tomography Measured Central Subfield Thickness From Baseline
Description: Change in central subfield thickness is followup central subfield retinal thickness minus baseline thickness.
Time Frame: Baseline to 6 Months
Measure: Median (Inter-Quartile Range); unit: microns
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
microns | -160 [-258 to -87]

3. Secondary Outcome: Surgical Complications From Baseline to Six Months
Description: Including intraoperative and perioperative medical complications. Same subject could have more than one complication
Time Frame: Baseline to 6 months
Measure: Number; unit: Participants
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
Participants
  Total | 16
  Vitreous hemorrhage | 5
  Additional vitreomacular interface abnormalities | 2
  Elevated intraocular pressure requiring treatment | 7
  Retinal Detachment | 3
  Endophthalmitis | 1
  Double vision | 2
  Lamella hole | 1
  Choroidal effusion | 1
  Other | 2

4. Primary Outcome: Percent of Participants With Change in Visual Acuity From Baseline to Six Months
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
Percentage of Participants
  Percent with 10 or more letter imporvement | 38 [28 to 49]
  Percent with 10 or more letters worsening | 22 [13 to 31]

5. Primary Outcome: Change in Optical Coherence Tomography Central Subfield Thickness From Baseline to 6 Months
Description: Change in thickness is followup thickness minus baseline thickness.
Time Frame: Baseline to 6 months
Measure: Number; unit: participants
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Number analyzed (Participants) | 87
participants
  Central subfield decrease of 100 microns or more | 49
  Central subfield decrease of 50 microns or more | 61
  Central subfield increase of 50 microns or more | 3
  Central subfield thickening decrease of >=50% | 50
  Central subfield less than 250 microns at 6 months | 33

ADVERSE EVENTS:
Arm/Group | Diabetic Macular Edema and Vitreomacular Traction
Serious Adverse Events (participants affected / at risk) | 4/87
Other Adverse Events (participants affected / at risk) | 12/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetic Macular Edema and Vitreomacular Traction (N=87)
retinal detachment (Eye disorders) | 3
Endophthalmitis (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetic Macular Edema and Vitreomacular Traction (N=87)
Vitreous haemorrhage (Eye disorders) | 5
Additional vitreomacular interface abnormalities (Eye disorders) | 2
Elevated intraocular pressure requirering treatment (Eye disorders) | 7
Double Vision (Eye disorders) | 2
Lamella hole (Eye disorders) | 1
Choroidal effusion (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No